CLINICAL TRIAL: NCT02728375
Title: Innovative Game-Based Rehabilitation Platform for Children With Motor and Cognitive Impairments Due to Neuro-developmental Disorders and Acquired Brain Injuries
Brief Title: Game-Based Rehabilitation Platform for Children With Neurodevelopmental Disorders and Acquired Brain Injuries
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Manitoba (Other)
Collaborators: SDM College of Physiotherapy (Other); Christian Medical College and Hospital, Ludhiana, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H2016:061
Record Dates: First submitted 2016-03-22; First posted 2016-04-05 (Estimated); Last update posted 2016-04-05 (Estimated); Status verified 2016-03

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Computer gaming hand exercise regimen (Experimental): Computer gaming hand exercise regimen using common objects of daily life. The hand exercises are coupled with commercially available computer games and will be performed 45 minutes,three times per week for sixteen weeks
  Interventions: Other: computer game based rehabilitation protocol
- Conventional hand exercise program (Active Comparator): Exercises targeted to improve finger range of motion and hand strength. The exercises will be performed 45 minutes, three times per week for sixteen weeks
  Interventions: Other: Conventional therapy protocol

INTERVENTIONS:
Other: computer game based rehabilitation protocol — Participants who consent to take part in the study will be asked to use objects instrumented with the miniature motion mouse to play various therapeutic yet entertaining games while handling and moving the test therapeutic objects as a part of experimental therapy protocol. The objects used will be everyday items; a) lifting/rotating a sports ball small beach ball which requires bimanual handling, b) rolling a cylinder object (diameter 6-10 cm with fingers extended and using elbow and shoulder motion, c) grasping grasp small glass and then a sponge ball with whole hand and rotating (supination- pronation motion) d) motion of a small wand (pencil) with 3-finger pinch grip and using hand-wrist motion, and e) turning of a key with 2-finger pinch fine finger control. These objects represent a wide range of physical properties requiring different modes of manipulation and functional demands sufficient to test the assessment tool.
  Arms: Computer gaming hand exercise regimen
Other: Conventional therapy protocol — In control group: 1) Stretching of Biceps, Lattisimusdorsi, Pronators, Thumb muscles. 2) Weight Bearing Exercises. 3) CIMT for 20 min per day for 3-4 weeks, repeat each task 15-20 times. Pegboard activities, Rings: reaching- removing and putting back, Ball throw (under and over arm) - at basket which is kept 10 to 15 meter distance, opening bottle cap (large size bottle), Opening and closing door handle activity, Holding water bottle, bag in hand and transfer to 10 to 20 meter distance, Crumbling paper, Clay activities, Picking marbles from sand 4)Hand arm bimanual activities: Throwing ball with both hands, Holding ball with both hands and transfer, Holding bolster and keeping at place, Holding notebook in both hands, Holding rack with both hands, Holding plate in one hand and spoon in other hand, Pushing door or wall both hands.
  Arms: Conventional hand exercise program

SUMMARY:
This research project focuses on the evaluation of an engaging exercise and cognitive computer game-based platform and embedded assessment tools for use in clinical practice and its transition to use in the home, and elementary classrooms. The goal of our research program is to produce innovative therapeutic point-of-care and cost-effective delivery system leading to better long-term health outcomes for toddlers and children with neurodevelopmental disabilities. The program is grounded on our technological developments and on current research documenting the benefits of computer-aided learning tools, exercise gaming applications in rehabilitation and principles of adaptive learning and neuroplasticity. We will conduct a randomized controlled trial to study the feasibility and effectiveness of a computer-aided, game-based repetitive task practice (RTP) program designed for training of fine and gross motor skills of the hand-arms and psychomotor skills (which) in young children with CP.

DETAILED DESCRIPTION:
This research project focuses on the evaluation of an innovative, engaging computer game-based exercise system for use in rehabilitation of young children with cerebral palsy, and its transition for use in home. The goal of this research program is to produce high quality therapeutic point-of-care approaches and cost-effective delivery systems leading to better long-term health outcomes. At present, the challenges entailed in providing therapy services continue to put identified children at risk of missing opportunities to maximize their neuro-developmental capacities, sustain any behavioral recovery and prevent future complications.

Canada and India face a growing population of children with neuro-developmental disabilities distributed across broad geographic regions. Cerebral palsy is the most common neuro-developmental disability in childhood. The prevalence of cerebral palsy (CP) in developing countries is estimated to be 5 to 10 times greater than in North America. Children with CP can result in deficits in fine and gross motor skills and often have co-occurring deficits in attention and cognitive functions. Half of these children with CP have impaired upper extremity function (reaching, grasping and manipulating objects). The ability to perform functional tasks with the upper extremities is an important predictor of success in daily activities and participation in school, leisure and other aspects of community life.

There are many things to consider when developing therapy programs designed to improve motor and psychomotor skills for affected children to maximize their neuro-developmental capacities and to prevent the development of secondary disabilities. Intense repetitive task practice such as, constraint-induced movement therapy is one of the few effective neuro-rehabilitative strategies shown to improve upper extremity motor function in children with CP, with potential to overcome developmental difficulties. Constraint induced movement therapy consists of constraining the use of the unaffected upper limb to encourage use of the affected upper limb. However it is often difficult to engage children in therapy and sustain motivation to engage in intense repetitive task practice in using the affected upper limb. Thus, there is a need for effective approaches and tools that motivate young children with CP to complete long-term neuro-rehabilitation programs and to provide developmental opportunities.

Digital media and gaming have received considerable interest from researchers and clinicians as a model for learning a broad range of complex tasks and facilitating the transfer of skills to daily life. These emerging rehabilitation technologies have the potential to improve clinical outcomes and child participation because they are engaging, motivating and now accessible. For this purpose investigators have developed a computer game-based rehabilitation and learning platform (CRP). This approach combines fine and gross motor exercises and cognitive activities appropriate for children with neuro- developmental disorders. The approach is designed to provide engaging, high-quality, personalized therapy in the clinical rehabilitation setting, and which could also be implemented in the school and home via Tele rehabilitation.

Research Goal:

This research project focuses on the evaluation of an engaging exercise and cognitive computer game-based platform and embedded assessment tools for use in clinical practice and its transition to use in the home, and elementary classrooms. The goal of this research program is to produce innovative therapeutic point-of-care and cost-effective delivery system leading to better long-term health outcomes for toddlers and children with neurodevelopmental disabilities. The program is grounded on investigators technological developments and on current research documenting the benefits of computer-aided learning tools, exercise gaming applications in rehabilitation and principles of adaptive learning and neuroplasticity. Investigators will conduct a randomized controlled trial to study the feasibility and effectiveness of a computer-aided, game-based repetitive task practice (RTP) program designed for training of fine and gross motor skills of the hand-arms and psychomotor skills (which) in young children with CP.

RESEARCH PROJECT OBJECTIVE 1

The CRP includes a designed rehabilitation assessment game which is capable of monitoring every child's performance during therapy. It quantifies motor skill parameters, as well as, visual-spatial skills and executive cognitive functions. It produces electronic records for these outcome measures and thus allows us to track change over time. It also provides timely feedback to child and therapist.

Objective: To evaluate the test-retest reliability and convergent validity of the assessment tool embedded in the game-based rehabilitation platform. Specifically for fine and gross motor skills and psychomotor skills in children aged 4-11 years (n= 40) diagnosed with cerebral palsy or acquired brain injuries. The new tool will be compared to commonly used outcome measures i.e. Quality of Upper Extremity skills test (QUEST) and Peabody Developmental Motor Scale version 2 (PDMS-2). This will provide a reliable test protocol and valid measures that can accurately and quickly quantify hand-arm function independent of object-task type, for use in daily clinical practice and research. Two common tests of fine and gross motor skill in CP children; a) Quality of Upper Extremity Skills Test (QUEST) and b) Peabody Developmental Motor Scale-2. We hypothesized that the performance measures of the game-based assessment tool would:

1. Exhibit high test retest reliability (Intra class correlations >0.7), and Standard error of measures less than 20% of the group mean
2. Show moderate convergent validity (correlations, r>0.06) with the primary outcome measures.

RESEARCH PROJECT OBJECTIVE 2

An exploratory randomized clinical trial will be conducted to evaluate the feasibility and benefits of the game-based rehabilitation program on fine manual dexterity skills and gross motor skills in children aged 4-11 years (n= 60) diagnosed with cerebral palsy. Two groups of children will be examined, one group will receive the experimental game-based program and the other group will receive usual therapy. Each program would take 16 weeks, three therapy sessions per week. Using a process of randomization, participants will be assigned to either experimental or control group after the initial assessment and screening performed by a blind assessor. Before the treatment sessions begin, after the end of 16 weeks and during a follow up session after 16 weeks, a clinician will conduct regular assessment sessions with the participant to mark the progress till date.

Investigators will be examining the feasibility of assessment tool embedded in the game-based rehabilitation platform and also the usability safety and appeal of the protocol. Investigators will observe a estimation of effectiveness on this sample using mixed method Analysis of Variance for within (repeated measure) and between group effects.

STUDY DESIGN: Exploratory Randomized Clinical Trial

METHOD OF COLLECTION OF DATA:

Ethical clearance for the study has been obtained from the Institutional Ethical Committee of S. D. M. College of Medical Sciences and Hospital, Dharwad and will be obtained from Institutional Ethical committee of Christian Medical College, Ludhiana, India. Participants will be recruited by clinicians working in Outpatient Department, S.D.M. Hospital, Dharwad, India and Christian Medical College and Hospital, Ludhiana, India. Participants who consent to take part in the study will be asked to use objects instrumented with the miniature motion mouse to play various therapeutic yet entertaining games while handling and moving the test therapeutic objects as a part of experimental therapy protocol. The objects used will be everyday items; a) lifting/rotating a sports ball small beach ball which requires bimanual handling, b) rolling a cylinder object (diameter 6-10 cm with fingers extended and using elbow and shoulder motion, c) grasping grasp small glass and then a sponge ball with whole hand and rotating (supination- pronation motion) d) motion of a small wand (pencil) with 3-finger pinch grip and using hand-wrist motion, and e) turning of a key with 2-finger pinch fine finger control. These objects represent a wide range of physical properties requiring different modes of manipulation and functional demands sufficient to test the assessment tool. In control group: 1) Stretching of Biceps, Lattisimus dorsi, Pronators, Thumb muscles. 2) Weight Bearing Exercises. 3) CIMT for 20 min per day for 3-4 weeks, repeat each task 15-20 times. Pegboard activities, Rings: reaching- removing and putting back, Ball throw (under and over arm) - at basket which is kept 10 to 15 meter distance, opening bottle cap (large size bottle), Opening and closing door handle activity, Holding water bottle, bag in hand and transfer to 10 to 20 meter distance, Crumbling paper, Clay activities, Picking marbles from sand 4)Hand arm bimanual activities: Throwing ball with both hands, Holding ball with both hands and transfer, Holding bolster and keeping at place, Holding notebook in both hands, Holding rack with both hands, Holding plate in one hand and spoon in other hand, Pushing door or wall both hands.

Further if parents have any queries regarding the study they can report to the principal investigators. The parents would be reassured that information would be kept confidential and will be used only for study purpose.

ELIGIBILITY:
Inclusion Criteria:

* Children with Cerebral Palsy
* Age between 4-11 years
* Moderate upper extremity impairments and fine motor control abnormalities along with mild-moderate cognitive impairment.

Exclusion Criteria:

* Child with visual impairment.
* Auditory impairment
* Orthopedic conditions such as recent fractures, fixed deformities of upper limb
* Any surgical intervention 6 months before the study or who intended to receive within the period of study.
* Non willing parents.

Tools For screening:

1. Manual Ability Classification System (MACS) (Scores: Level 2, 3 and 4)
2. Gross Motor Function Classification Scale (GMFCS) (Scores: Level 2, 3 and 4)
3. Mini mental state examination scale for Children (23 and above out of 30)
4. Ashworth scale for spasticity of hand and arm (Level 1, 1+, 2)

Ages: 4 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2016-10 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Quality of Upper Extremity Skills Test | Change from baseline at 16 weeks and 6 months.
Peabody Developmental Motor Scale- 2 Fine motor Quotient | Change from baseline at 16 weeks and 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Szturm, Ph.D., Principal Investigator — Associate Professor
Locations (1):
- University of Manitoba, Winnipeg, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kanitkar A, Parmar ST, Szturm TJ, Restall G, Rempel G, Sepehri N. Parents' Perspectives on a Computer Game-Assisted Rehabilitation Program for Manual Dexterity in Children With Cerebral Palsy: Qualitative Analysis of Expectations, Child Engagement, and Benefits. JMIR Rehabil Assist Technol. 2021 May 31;8(2):e24337. doi: 10.2196/24337. PMID 34057424
- [Derived] Kanitkar A, Szturm T, Parmar S, Gandhi DB, Rempel GR, Restall G, Sharma M, Narayan A, Pandian J, Naik N, Savadatti RR, Kamate MA. The Effectiveness of a Computer Game-Based Rehabilitation Platform for Children With Cerebral Palsy: Protocol for a Randomized Clinical Trial. JMIR Res Protoc. 2017 May 18;6(5):e93. doi: 10.2196/resprot.6846. PMID 28526673